CLINICAL TRIAL: NCT02120781
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Azficel-T for the Treatment of Vocal Fold Scarring and Age-Related Dysphonia
Brief Title: Controlled Study to Evaluate the Safety and Efficacy of Azficel-T for Vocal Fold Scarring and Age-Related Dysphonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FI-V-002
Record Dates: First submitted 2014-03-21; First posted 2014-04-23 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Dysphonia Resulting From Vocal Fold Scarring; Age-related Dysphonia
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azficel-T (autologous fibroblasts) (Experimental): Azficel-T will be injected into the vocal fold(s) three times at two week intervals.
  Interventions: Biological: Azficel-T (autologous fibroblasts)
- Control (Placebo Comparator): Sterile saline will be injected into the vocal fold(s) three times at two week intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Azficel-T (autologous fibroblasts) — Autologous fibroblasts will be cultured from three 3-mm post auricular punch biopsies. Biopsies will be shipped from the clinical sites to the Fibrocell manufacturing site where the cells will be harvested, tested for sterility, endotoxin level, cell identity, viability and concentration. When the desired cell number is reached, cells will be transported to the investigative site as a suspension in shipping media.
  Depending upon the clinical circumstances for each subject, the vocal fold(s) will be injected transorally or percutaneously in order to deposit 1.0 mL of study drug into the lamina propria layer of each vocal fold. The injection process will be visualized via a flexible fiberoptic laryngoscope inserted through the nostril.
  Other Names: LAVIV™
  Arms: Azficel-T (autologous fibroblasts)
Drug: Placebo — Subjects randomized to placebo will receive injections of sterile saline into the vocal fold(s).
  Other Names: Sterile saline for injection
  Arms: Control

SUMMARY:
The objectives of this study are to assess the safety of azficel-T treatment for dysphonia related to vocal fold function and to evaluate the efficacy of azficel-T for the treatment of dysphonia related to vocal fold function.

DETAILED DESCRIPTION:
Twenty subjects with dysphonia caused by vocal fold scarring or age-related dysphonia will be randomized for treatment with autologous cultured fibroblasts (azficel-T, n=14) or placebo (saline, n=6). Subjects will receive treatment to the vocal fold(s) in the lamina propria compartment.

Subjects with both unilateral and bilateral vocal fold scarring will be treated in this study. Only one vocal fold will be treated at each treatment session alternating to the opposite vocal fold (if applicable) at the next treatment. Subjects are to receive a total of three treatments with study drug (azficel-T or placebo) if one vocal fold is to be treated and up to a total of six treatments with study drug (azficel-T or placebo) if two vocal folds are to be treated at approximately 2-week intervals. Follow-up examinations will be performed at 1, 4, 8, and 12 months after the final treatment. If there are any evident safety issues, follow-up treatments will be delayed or withheld.

In the Blinded Phase of the study, subjects will be followed for safety and efficacy for 4 months after the final treatment. After all subjects have completed the 4-month follow-up visit, the study will be unblinded and subjects will continue to be followed for safety for 12 months after the final treatment. Efficacy assessments will be made through the 12-month follow-up visit in order to document any duration of effect. All AEs that have an onset date from biopsy through the 4-month follow-up visit will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read and signed the Institutional Review Board (IRB)-approved informed consent form (ICF) before treatment
2. Subject is at least 18 years of age
3. Subject has presence of unilateral or bilateral vocal fold scarring or age-related dysphonia, as diagnosed by medical history and physical examination
4. Subject must have Grade 1-2 mucosal waves as determined by videostroboscopy
5. Subject has failed any one or more of the following treatments including, but not limited to, anti-reflux regimen, speech therapy, or vocal fold injection augmentation prior to screening
6. Subject feels that their voice quality is a major handicap
7. Subject must have a blood sample tested and found to be non-reactive for human immunodeficiency virus-1 (HIV-1) antibody, hepatitis B surface antigen and hepatitis C virus (HCV) antibody
8. If the subject is female and of childbearing potential, she must agree to use a medically acceptable means of birth control, and test negative on a urine pregnancy test
9. Subject must be willing and able to follow study procedures and instructions

Exclusion Criteria:

1. Subject is pregnant or lactating
2. Subject is a smoker
3. Subject has an upper respiratory infection at baseline (subject can be rescheduled after four weeks)
4. Subject is already participating, or has participated in another clinical trial involving therapeutic intervention within 30 days prior to enrollment
5. Subject plans to begin or continue other vocal fold therapies during the course of this study
6. Subject has other concurrent laryngeal pathology including lesions that would require removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Chhetri, MD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - Surgery/Head and Neck, David Geffen School of Medicine at UCLA, Los Angeles, California
  - Dept of Otolaryngology, Stanford Univ Medical Center, Stanford, California
  - NYU Langone Medical Center, New York, New York

REFERENCES:
- [Background] Chhetri DK, Berke GS. Injection of cultured autologous fibroblasts for human vocal fold scars. Laryngoscope. 2011 Apr;121(4):785-92. doi: 10.1002/lary.21417. Epub 2011 Feb 1. PMID 21287562

RESULTS

PARTICIPANT FLOW:
Groups:
- Azficel-T (Autologous Fibroblasts): Azficel-T will be injected into the vocal fold(s) three times at two week intervals.
  Azficel-T (autologous fibroblasts): Autologous fibroblasts will be cultured from three 3-mm post auricular punch biopsies. Biopsies will be shipped from the clinical sites to the Fibrocell manufacturing site where the cells will be harvested, tested for sterility, endotoxin level, cell identity, viability and concentration. When the desired cell number is reached, cells will be transported to the investigative site as a suspension in shipping media.
  Depending upon the clinical circumstances for each subject, the vocal fold(s) will be injected transorally or percutaneously in order to deposit 1.0 mL of study drug into the lamina propria layer of each vocal fold. The injection process will be visualized via a flexible fiberoptic laryngoscope inserted through the nostril.
Period: Overall Study
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Started | 15 | 6
Completed | 11 | 5
Not Completed | 4 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Completion not documented | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (13.95) | 68.3 (19.37) | 63.7 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 5 | 18
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Improvement From Baseline in Mucosal Wave Grade
Description: Any improvement from baseline in mucosal wave grade using videostrobscopy to assess the pliability of vocal folds which is visualized as mucosal waves on the vocal fold surface while a participant is phonating a sustained vowel sound.
Time Frame: Four months after final treatment, or up to a total of 25 weeks from baseline with unilateral treatment and 27 weeks from baseline for bilateral treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 14 | 5

2. Primary Outcome: Number of Participants With an Absolute Change in Voice Handicap Index Score (Decrease of 18 or More Points) From Baseline
Description: Absolute change (decrease by 18 or more points) from baseline in the Voice Handicap Index (VHI) score 4 months after the final treatment.
  The VHI is a 30-item test with 10 items in 3 subscales: emotional, physical, and functional. Each item is scored on a 5-point scale: "0" indicating the subject never felt this about the voice problem and "4" indicating the subject always felt this to be the case. An 8-point difference on any subscale (sub-scale range 0-40, higher values represent worse outcomes) has been found to be significant, as was an 18-point difference in the total VHI score (Total scale range 0-120, higher values represent worse outcomes).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 4 | 3

3. Primary Outcome: Mean Percentage Change From Baseline in Voice Handicap Index Score
Description: Mean percentage change from baseline in the Voice Handicap Index (VHI) score 4 months after the final treatment. The VHI is a 30-item test with 10 items in 3 subscales: emotional, physical, and functional. Each item is scored on a 5-point scale: "0" indicating the subject never felt this about the voice problem and "4" indicating the subject always felt this to be the case. An 8-point difference on any subscale (sub-scale range 0-40, higher values represent worse outcomes) has been found to be significant, as was an 18-point difference in the total VHI score (Total scale range 0-120, higher values represent worse outcomes).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
percentage of change | -10.00 (57.074) | -28.86 (51.949)

4. Primary Outcome: Number of Participants With at Least One Level of Improvement in Perceptual Analysis of Dysphonia Using GRBAS Scale.
Description: Perceptual analysis of dysphonia using the Grade of Dysphonia, Roughness, Breathiness, Asthenia, Strain (GRBAS) scale is assessed by a blinded voice clinician 4 months after the final treatment. The voice clinician considers pre- and post-treatment voice recordings, and categorizes the individual parameters on the GRBAS scale (absent, mild, moderate, and severe). Scores of mild, moderate, or severe represent increasingly worse outcomes than a score of absent.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 4 | 2

5. Primary Outcome: Number of Participants With at Least One Level of Improvement in Perceptual Analysis of Roughness Using GRBAS Scale.
Description: Perceptual analysis of roughness using the Grade of Dysphonia, Roughness, Breathiness, Asthenia, Strain (GRBAS) scale is assessed by a blinded voice clinician 4 months after the final treatment. The voice clinician considers pre- and post-treatment voice recordings, and categorizes the individual parameters on the GRBAS scale (absent, mild, moderate, and severe). Scores of mild, moderate, or severe represent increasingly worse outcomes than a score of absent.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 1 | 2

6. Primary Outcome: Number of Participants With at Least One Level of Improvement in Perceptual Analysis of Breathiness Using GRBAS Scale.
Description: Perceptual analysis of breathiness using the Grade of Dysphonia, Roughness, Breathiness, Asthenia, Strain (GRBAS) scale is assessed by a blinded voice clinician 4 months after the final treatment. The voice clinician considers pre- and post-treatment voice recordings, and categorizes the individual parameters on the GRBAS scale (absent, mild, moderate, and severe). Scores of mild, moderate, or severe represent increasingly worse outcomes than a score of absent.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 5 | 0

7. Primary Outcome: Number of Participants With at Least One Level of Improvement in Perceptual Analysis of Asthenia Using GRBAS Scale.
Description: Perceptual analysis of asthenia using the Grade of Dysphonia, Roughness, Breathiness, Asthenia, Strain (GRBAS) scale is assessed by a blinded voice clinician 4 months after the final treatment. The voice clinician considers pre- and post-treatment voice recordings, and categorizes the individual parameters on the GRBAS scale (absent, mild, moderate, and severe). Scores of mild, moderate, or severe represent increasingly worse outcomes than a score of absent.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 4 | 3

8. Primary Outcome: Number of Participants With at Least One Level of Improvement in Perceptual Analysis of Strain Using GRBAS Scale.
Description: Perceptual analysis of strain using the Grade of Dysphonia, Roughness, Breathiness, Asthenia, Strain (GRBAS) scale is assessed by a blinded voice clinician 4 months after the final treatment. The voice clinician considers pre- and post-treatment voice recordings, and categorizes the individual parameters on the GRBAS scale (absent, mild, moderate, and severe). Scores of mild, moderate, or severe represent increasingly worse outcomes than a score of absent.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
Number analyzed (Participants) | 15 | 6
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 months after the first study treatment.
Arm/Group | Azficel-T (Autologous Fibroblasts) | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/6
Other Adverse Events (participants affected / at risk) | 13/15 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azficel-T (Autologous Fibroblasts) (N=15) | Control (N=6)
intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azficel-T (Autologous Fibroblasts) (N=15) | Control (N=6)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
laryngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
laryngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
laryngitis (Infections and infestations) | 1 (1) | 1 (1)
bronchitis (Infections and infestations) | 0 (0) | 1 (1)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
hordeolum (Infections and infestations) | 1 (2) | 0 (0)
post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
sinusitis (Infections and infestations) | 0 (0) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
injection site pain (General disorders) | 0 (0) | 1 (1)
injection site paraesthesia (General disorders) | 1 (1) | 0 (0)
procedural anxiety (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
blood urine present (Investigations) | 1 (1) | 0 (0)
hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
restless leg syndrome (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No